CLINICAL TRIAL: NCT06303050
Title: Additional Effects of Mental Imagery Along With Task Oriented Training on Kinesiophobia in Patients With Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Urooj Amir
Record Dates: First submitted 2024-03-04; First posted 2024-03-12 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Stroke, Cardiovascular
Keywords: Mental Imagery; Kinesiophobia; Task oriented training
MeSH Terms: conditions — Myocardial Infarction; Kinesiophobia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mental Imagery with task Oriented training group (Experimental): Participants will perform warm-up exercise for 5 minutes to prepare the body for functional task and to improve overall performance.
  Interventions: Other: Mental Imagery with task Oriented training group
- Task Oriented training group (Active Comparator): Task oriented training In standing, forward stepping and sideward stepping, reaching in standing, Transition from sit to stand, Walk then back to sit, Walk with even steps, Walk with carrying objects.
  Interventions: Other: Task Oriented training group

INTERVENTIONS:
Other: Mental Imagery with task Oriented training group — Study will be conducted after the approval of Ethical review board. After the initial evaluation will be done on participants underlying eligibility criteria. The experimental group will receive 20 minutes of MI training followed by 25 minutes of TOT for a total of 45 minutes, 5 days per week for 6 weeks. During each 45 minutes of session, the participants will perform warm-up exercise for 5 minutes to prepare the body for functional task and to improve overall performance. Regular breaks will give to the participants to avoid overexertion and fatigue during 45 minutes of continues practice. The 2 minutes rest period will provide to the partici-pants during each practice session
  Arms: Mental Imagery with task Oriented training group
Other: Task Oriented training group — Study will be conducted after the approval of Ethical review board. After the initial evaluation will be done on participants underlying eligibility criteria. The control group will receive the Task oriented training for 25-30 minutes, 05 days a week for 06 weeks consisting of Warm up Period, Task oriented training In standing, forward stepping and sideward stepping, reaching in standing, Transition from sit to stand, Walk then back to sit, Walk with even steps, Walk with carrying objects.
  Arms: Task Oriented training group

SUMMARY:
The objective of this study to determine the effect of mental imagery and task oriented training on Kinesiophobia in stroke patients. And to determine the association of Kinesiophobia with gait and balance in stroke patients. Patients will be divided into experimental and control group. Randomized participants will be allocated into control and experimental group. The experimental group will receive 20 minutes of MI training followed by 25 minutes of TOT for a total of 45 minutes, 5 days per week for 6 weeks.

DETAILED DESCRIPTION:
Cerebrovascular accident (CVA),commonly known as stroke , occurs when blood flow to the brain is disrupted , either by a clot or by rupture in a blood vessel .It can lead to severe neurological damaged or even death. A stroke can cause neurological deficits in various domains of brain areas, include motor, sensory/perceptive, visual, language, intelligence and emotion. Motor deficits are one of the most common and disabling consequences of stroke.

Kinesiophobia is a psychological condition characterized by an excessive, irrational fear of movement and physical activity due to the belief that it will increase pain or worsen a pre medical condition. It can be a common obstacle to rehabilitation and recovery for individuals with various musculoskeletal or neurological conditions, including stroke.

MI has been recognized as an effective adjunct therapy to physical rehabilitation for various neurological conditions, including stroke. Task-oriented training is a widely adopted approach in stroke rehabilitation, which emphasizes the practice of functional tasks to promote motor skill learning and improve motor function.

However the potential benefits of combining mental imagery with task-oriented train-ing have not been fully explored. Therefore studying the additional effects of mental imagery along with task-oriented training on Kinesiophobia in patients with stroke is important for developing more effective and comprehensive rehabilitation interven-tions for stroke populations.

ELIGIBILITY:
Inclusion Criteria:

* Hemiplegic stroke patients
* Age above 45
* Both genders
* Patients having score >17 on Tempa Scale of Kinesiophobia
* Patients of score >21 on Berg Balance Scale

Exclusion Criteria:

* • Communication deficits and unable to follow instructions

  * A history of serious or unstable cardiac condition
  * Severe musculoskeletal problem and unable to stand or walk
  * History of other neurological diseases or unilateral neglect

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2023-12-07 (Actual); Primary Completion 2024-06-07 (Actual); Study Completion 2024-06-07 (Actual)

PRIMARY OUTCOMES:
Berg And Balance scale | 6 weeks
  changes from the baseline, Berg balance scale (BBS) is used for assessment of balance and fall risk, Higher scores on the BBS indicate greater independence and better ability to balance. In contrast, lower scores indicate a greater fall risk Items DESCRIPTION SCORE (0-4) Sitting to standing, Standing unsupported, Sitting unsupported, Standing to sitting, Transfers , Standing with eyes closed , Standing with feet together, Reaching forward with outstretched arm, Retrieving object from floor, Turning to look behind, Turning 360 degrees, Placing alternate foot on stool, Standing with one foot in front, Standing on one foot, TOTAL __/56
Tempa scale for kinesiophobia | 6 weeks
  It consists of 17 items asking patients to rate their responses to statements related to fear of movement and re injury. It has been widely used among patients with various types of pain and has been translated into several languages. The TSK-17 is a useful tool for assessing kinesiophobia and can aid clinicians in developing appropriate treatment plans for patients who may have fear of movement due to pain or injury (20). The TSK exhibit high level of in- ternal consistency across all items and is positively associated with related measures of fear avoidance, pain catastrophizing, pain related disability. In the Finnish version of TSK the test-retest reliability
Ten-meter walk test | 6 weeks
  The 10- meter walk test is a commonly used tool to measure gait and walking speed in individuals with mobility impairments, including post-stroke individuals. During the test subjects are instructed to walk along a 10-meter walkway at their preferred walking speed, with or without a customary walking device, without any break to the end point. The time taken to recover the middle 4 meters of the walkway is recorded to obtain a rhythmic phase of walking speed. This ensures that the acceleration and deceleration phases of walking are excluded from the measurement of walking speed. Then the time required over three trials is converted to walking speed by dividing the distance (6 meters) by the time taken in seconds to complete the walk.
Dynamic gate index | 6 weeks
  The DGI tests the ability of the participant to maintain walking balance while responding to different task demands, through various dynamic conditions.
  It includes eight items, walking on level surfaces, changing speeds, head turns in horizontal and vertical directions, walking and turning 180 degrees to stop, stepping over and around obstacles, and stair ascent and descent.
  Each item is scored on a scale of 0 to 3, with 3 indicating normal performance and 0 representing severe impairment. The best possible score on the DGI is a 24.
Time Up and Go Test | 6 weeks
  Timed up and go test is used for the assessment of falls risk among the elderly population. The Timed "Up and Go" (TUG) Test measures, in seconds, the time is taken by an individual to stand up from a standard armchair (approximate seat height of 46 cm, arm height 65 cm), walk a distance of 3 meters (approximately 10 feet), turn, walk back to the chair, and sit down. Normal healthy elderly usually complete the task in 10 seconds or less. Very frail or weak elderly with poor mobility may take 2 minutes or more. Clinical guide: <10 seconds = normal <20 seconds = good mobility, can go out alone, mobile without a gait aid <30 seconds = problems, cannot go outside alone, requires a gait aid A score of more than or equal to 14 seconds has been shown to indicate a high risk of falls.

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Azhar, MS-NMPT, Principal Investigator — Riphah International University
Locations (1):
- Khyber Medical University, Peshawar, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No